CLINICAL TRIAL: NCT00942344
Title: An 8-week, Multicenter, Randomized, Double-blind, Factorial Phase II Study to Evaluate Dose-response Relationship of Amlodipine and Losartan Combination in Patients With Essential Hypertension.
Brief Title: Efficacy and Safety of Amlodipine and Losartan in Patients With Essential Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Director, Hanmi Pharmaceutical Company Limited
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: HM-ALOS-201
Record Dates: First submitted 2009-07-17; First posted 2009-07-20 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
Keywords: Amlodipine; Losartan; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Amlodipine plus Losartan — amlodipine/losartan 5/50mg, 5/100mg, 10/50mg, 10/100mg
  Other Names: Amosartan
Drug: Amlodipine — amlodipine 5mg, 10mg
Drug: Losartan — Losartan 50mg, 100mg

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of fixed combination of amlodipine(5mg or 10mg) and losartan (50 mg or 100 mg), amlodipine and losartan alone in reducing blood pressure. The study will investigate the dose response relationship for the combinations and monotherapies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75
* Patients with essential hypertension {95 mmHg ≤ sitDBP< 115 mmHg at the end of placebo run-in treatment period}

Exclusion Criteria:

* Patients with mean sitSBP ≥ 200 mmHg
* Patients with known hypersensitivity to Dihydropyridine or angiotensin II receptor blockers
* Patients with secondary hypertension or suspected secondary hypertension
* Patients with malignant hypertension
* Patients who have received any medications with possible interactions with study drugs
* Patients with uncontrolled diabetes
* Patients with severe heart disease or severe cerebrovascular disease
* Patients with clinically significant hematological test results, renal disease (serum creatinine) or liver disease (ALT or AST)
* Patients with a history of malignant disease
* Patients with a history of autoimmune disease
* Women with a positive pregnancy test result, breast feeding or intention of pregnancy during the trial
* Patients inappropriate to be included in study population due to other reasons at the discretion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2007-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Average changes from baseline in sitDBP | Week 8

SECONDARY OUTCOMES:
Average changes from baseline in sitDBP | Week 4
Average changes from baseline in sitSBP | Week 4, 8
Blood pressure responder rate | Week 4, 8

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Yun Cho, M.D., Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- 14 sites in Korea, Seoul, Busan, Etc., South Korea

REFERENCES:
- [Derived] Park CG, Youn HJ, Chae SC, Yang JY, Kim MH, Hong TJ, Kim CH, Kim JJ, Hong BK, Jeong JW, Park SH, Kwan J, Choi YJ, Cho SY. Evaluation of the dose-response relationship of amlodipine and losartan combination in patients with essential hypertension: an 8-week, randomized, double-blind, factorial, phase II, multicenter study. Am J Cardiovasc Drugs. 2012 Feb 1;12(1):35-47. doi: 10.2165/11597170-000000000-00000. PMID 22217192